CLINICAL TRIAL: NCT02212782
Title: A Randomized, Open-label, Multiple-dose, Crossover Phase I Clinical Study to Evaluate DW1029M Influence the Pharmacokinetic Profiles of Linagliptin After Oral Administration in Healthy Male Volunteer
Brief Title: the Pharmacokinetic Profiles of Linagliptin With DW1029M
Acronym: PLID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: DW1029M-I-6
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: Healthy
MeSH Terms: interventions — Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Group (Experimental): 1st oral administration of Linagliptin 5mg and 2nd oral administration of DW1029M 1200mg and Linagliptin 5mg
  Interventions: Drug: Linagliptin 5mg; Drug: DW1029M 1200mg and Linagliptin 5mg
- B Group (Experimental): 1st oral administration of DW1029M 1200mg and Linagliptin 5mg and 2nd oral administration of Linagliptin 5mg
  Interventions: Drug: Linagliptin 5mg; Drug: DW1029M 1200mg and Linagliptin 5mg

INTERVENTIONS:
Drug: Linagliptin 5mg — Linagliptin 5mg once daily for 7 days
  Other Names: Trajenta Tablet
Drug: DW1029M 1200mg and Linagliptin 5mg — Linagliptin 5mg 1 tablet once daily and DW1029M 300mg 2 tablets b.i.d for 7 days
  Other Names: Concomitant of DW1029M 1200mg and Linagliptin 5mg

SUMMARY:
Phase I clinical study to evaluate DW1029M influence the pharmacokinetic profiles of Linagliptin after oral administration in healthy male volunteer.

DETAILED DESCRIPTION:
A Randomized, open-label, multiple-dose, crossover phase I clinical study to evaluate DW1029M influence the pharmacokinetic profiles of Linagliptin after oral administration in healthy male volunteer.

ELIGIBILITY:
Inclusion Criteria:

* A healthy adult within the range of 19 to 55 years old at the time of screening
* Body Mass Index(BMI)=17.5~30.5kg/m2, one with weight of more than 55kg (BMI= kg/(m)2)
* Congenital or chronic diseases within the last three years, there is no medical examination results of popular characters with no psychotic symptoms or findings
* Doctor checks conducted hematology, blood chemistry, urinalysis and laboratory tests, including an electrocardiogram(EKG) performed during screening tests such as a suitable test subjects who judged
* The purpose of the test participants prior to testing, information, and to hear about the free will fully explain to participate in this study, according to the Institutional Review Board(IRB)-approved consent form signed by the parties in writing

Exclusion Criteria:

* one with clinically significant blood, kidneys, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurological or allergic disease (but ,except for untreated seasonal allergies of asymptomatic at the time of administration) with medical history or evidence
* one with gastrointestinal disease(Such as esophageal stricture or achalasia of the esophagus disease, Crohn disease) to affect drug absorption or surgery(but, excluding simple appendectomy or hernia surgery) with medical history
* Alanine Aminotransferase(ALT) or Aspartate Aminotransferase(AST) > 2 times the upper limit of the normal range
* Within 6 months, 210 g / week of alcohol in excess of a history of regular characters (beer (5%) 1 cup (250 mL) = 10 g, soju(20%) 1 cup (50 mL) = 8 g, Wine (12%) 1 cup (125 mL) = 12 g)
* Take part in other clinical trials within two months
* Systolic Blood Pressure(SBP) ≥ 140 mmHg or Diastolic Blood Pressure (DBP) ≥ 90 mmHg
* The great history of alcohol or drug abuse within 1 year
* Taking medication of drug-metabolizing enzymes that are known to significantly induce or inhibit within 30 days
* More than 20 cigarettes a day smoker
* Taking medication of a prescription drug or nonprescription within 10 days,
* Within two months the whole blood donation have, within one month of the apheresis donation have
* Participate in clinical trials to test drug administration and may be at increased risk due to interpretation of test results, or may interfere with severe supply / chronic medical or mental condition or abnormal laboratory test values in character
* Patient with hypersensitivity to investigational products or ingredients
* Patient with Type 1 Diabetes or Diabetic ketoacidosis
* Described lifestyle in this protocol can comply with or can not
* One with other investigator judge to unsuitable

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cmax and AUC | 1st day and 43rd day, 5th day and 47th day, 6th day and 48th day : Predose(0, morning), 7th day and 49th day : Predose(0), 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour
  Maximum of Concentration(Cmax), Area Under Plasma Concentration-Time Curve(AUC)

SECONDARY OUTCOMES:
Pharmacokinetic Profile of Plasma | 1st day and 43rd day, 5th day and 47th day, 6th day and 48th day : Predose(0, morning), 7th day and 49th day : Predose(0), 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour
  Maximum drug concentration time(Tmax), Half-time(t1/2), Apparent renal clearance(CL/F), Apparent volume of distribution(Vd/F), Fluctuation[(Css,max-Css,min)/Css,av], Swing[(Css,max-Css,min)/Css,min]

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, M.D, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabukdo, South Korea